CLINICAL TRIAL: NCT06216158
Title: A Randomized Phase III Trial Assessing Iberdomide Versus Iberdomide Plus Isatuximab Maintenance Therapy Post Autologous Hematopoietic Stem Cell Transplantation in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Iberdomide vs. Iberdomide Plus Isatuximab Maintenance Therapy Post ASCT in Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: KKS Netzwerk (Network); Wuerzburg University Hospital (Other); Sanofi (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Elias Mai, Principal Investigator, University of Heidelberg Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMMG-HD9/DSMM XVIII
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; isatuximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Iberdomide (Active Comparator): 36 months of oral iberdomide administration; In cycle 1, dexamethasone is added as pre-medication
  Interventions: Drug: Iberdomide; Drug: Dexamethasone
- Arm B: Iberdomide plus isatuximab (Experimental): 36 months of oral iberdomide plus subcutaneous isatuximab administration; In cycle 1, dexamethasone is added as pre-medication
  Interventions: Drug: Iberdomide; Drug: Isatuximab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Iberdomide — Iberdomide p.o. (0.75 mg, day 1-21 of each 29-days cycle)
Drug: Isatuximab — Isatuximab s.c. (1400 mg, cycle 1: day 1, 8, 15, 22; cycles 2-3: day 1 and 15; from C4: day 1)
  Other Names: Sarclisa
  Arms: Arm B: Iberdomide plus isatuximab
Drug: Dexamethasone — Dexamethasone p.o. or i.v. (20 mg, cycle 1 only: day 1, 8, 15, 22)

SUMMARY:
The goal of this clinical trial is to compare a maintenance therapy consisting of iberdomide and isatuximab with an iberdomide-only regimen. The trial is the subsequent maintenance therapy to GMMG-HD8/DSMM XIX trial for patients with newly-diagnosed multiple myeloma. Patients with newly-diagnosed multiple myeloma who underwent a similar quadruplet induction/consolidation therapy regimen followed by at least one ASCT can also be recruited. The main question it aims to answer is:

• Will the addition of isatuximab lead to decreased amounts of measurable myeloma cells in the bone marrow after two years?

DETAILED DESCRIPTION:
Prospective, multicentre, randomised, parallel group, open, phase III clinical trial for a maintenance therapy, for patients who underwent an induction therapy and autologous stem cell transplantation (ASCT) in the GMMG-HD8/DSMM XIX trial or a similar quadruplet induction/consolidation therapy regimen followed by at least one ASCT.

Investigational Medicinal Product: Iberdomid (oral), isatuximab (subcutaneous administration via a wearable injector system).

Randomisation will be performed centrally by GMMG/DSMM offices after verification of the eligibility of the patient. At the time of study inclusion, randomization will be performed into arm A (iberdomide) or arm B (iberdomide + isatuximab). Randomization will be stratified by centrally assessed MRD negativity status (yes vs. no vs. unknown); assessed by NGF from BMA; sensitivity of 10^-5; independent of standard IMWG response) and number of HDM/ASCT (single vs. tandem).

Patients randomized in arm A will receive 39 cycles of the drug iberdomide, a Cereblon E3 Ubiquitin Ligase Modulating Drug (CELMoD®) that shares structural similarities to the immunomodulatory compounds (IMiDs) such as thalidomide and lenalidomide. Each cycle will last for 29 days. Patients in arm B will receive the same the 39 cycles of iberdomide plus monoclonal anti-CD38 antibody isatuximab subcutaneously. In both arms, patients will receive 20 mg dexamethasone in cycle 1, on the same days as the isatuximab administration in Arm B. End of study will be after 36 months of the maintenance therapy.

There is one primary objective:

- Demonstration of superiority of iberdomide plus isatuximab compared to iberdomide with respect to bone marrow minimal residual disease (MRD) negativity rates (sensitivity 2x10^-6 via next-generation flow cytometry [NGF]) after two years of maintenance therapy.

There is one key secondary objective:

- PFS, defined as time from randomization to disease progression or death from any cause, whichever occurs first.

Further secondary objectives are:

* Rates of sustained MRD negativity (at sensitivity levels of 10-5 and 2x10^-6 via NGF from BMA) after 1, 2 and 3 years of maintenance therapy.
* Conversion from MRD positive to negative (at sensitivity levels of 10^-5 and 2x10^-6 via NGF from BMA).
* Rates of best overall response to treatment (BOR).
* Rates of partial response (PR), very good partial response (VGPR), complete response (CR) and stringent complete response (sCR).
* Time-to-next-treatment (TTNT).
* PFS on subsequent line of therapy.
* Overall survival (OS).
* Improvement of IMWG response categories (PR, VGPR, CR, sCR).
* Proportions of patients in both treatment arms maintaining BOR and CR from baseline.
* Assessment of quality-of-life (QoL) via the EORTC-QLQC30, EORTC-QLQMY20, and EQ-5D-5L questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Prior inclusion and treatment within the GMMG-HD8 / DSMM XIX trial OR
* Received a quadruplet induction/consolidation therapy that consists of a proteasome inhibitor (PI) and immunomodulatory drug (IMiD) [e.g., bortezomib, thalidomide and dexamethasone, or bortezomib, lenalidomide and dexamethasone] with an anti-CD38 monoclonal antibody (isatuximab or daratumumab)
* Post HDM/ASCT consolidation containing similar substances as induction therapy is permitted
* Induction and consolidation therapy should make up a total of at least 4 up to 6 cycles, with a maximum of 2 consolidation cycles post HDM/ASCT AND
* Received at least one cycle high dose melphalan therapy (HDM) and autologous stem cell transplantation (ASCT)
* At least Partial Response (PR) according to IMWG criteria at inclusion in the trial
* Age of at least 18 years at trial inclusion
* WHO performance status of 0, 1, or 2
* Negative pregnancy test at inclusion (women of childbearing potential)
* For all men and women of childbearing potential: patients must be willing and capable to use adequate contraception during the complete therapy
* Ability of patient to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Subjects with gastrointestinal disease that may significantly alter the absorption of iberdomide
* Patient has known hypersensitivity (or contraindication) to any of the components of study therapy that are not amenable to premedication with steroids or H1 blockers and that would prohibit further treatment with these agents (e.g. known intolerance or hypersensitivity to infused proteins products, sucrose, histidine, and polysorbate 80 as well as intolerance to arginine and Poloxamer 188)
* Patients with a history of serious allergic reaction to another immunomodulatory agent (thalidomide, lenalidomide, or pomalidomide)", as angioedema and severe dermatologic reactions, including Grade 4 rash and exfoliative or bullous rash
* Patients currently being treated with strong inhibitors or inducers of CYP3A4/5
* Systemic AL amyloidosis (except for localized AL amyloidosis limited to the skin or the bone marrow), plasma cell leukemia or polyneuropathy, organomegaly, endocrinopathy, monoclonal-protein and skin abnormalities or Waldenström macroglobulinemia.
* Previous systemic anti-myeloma treatment other than administered within the GMMG-HD8 / DSMM XIX trial or other than defined in the inclusion criteria above (including up to two cycles cycle high dose melphalan therapy (HDM) and autologous stem cell transplantation (ASCT). Local, consolidative radiotherapy for myeloma disease is permitted unless performed in case of progressive disease according to IMWG criteria
* Severe cardiac dysfunction (NYHA classification III-IV)
* Significant hepatic dysfunction (ASAT and/or ALAT ≥ 3 times normal level and/or serum bilirubin ≥ 1.5 times normal level if not due to hereditary abnormalities as Gilbert's disease), unless related to MM or HDM/ASCT.
* Patients with active or uncontrolled hepatitis B or C or detectable liver disease due to hepatitis B or C. In case of history of hepatitis B or C, it must be clarified whether it has been overcome and negative circulating HBV-DNA or HCV-RNA must be provided. Positive hepatitis B status may only be acceptable in absence of circulating HBV-DNA or signs of chronic or acute infection and if an adequate prophylaxis is being implemented during the course of the study. Prophylaxis for patients with history of hepatitis B or C should be set on a patient individual basis.
* HIV positivity
* Patients with active, uncontrolled infections
* Patients with severe renal insufficiency (Creatinine Clearance < 30ml/min) or requiring hemodialysis
* Patients with peripheral neuropathy or neuropathic pain, grade 2 or higher (as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE, version 5.0)
* Patients with a history of any active malignancy during the past 5 years with the exception of following malignancies after curative therapy: basal cell carcinoma of the skin, squamous cell skin carcinoma, stage 0 cervical carcinoma or any in situ malignancy. A history of an early stage malignancy during the past 5 years may be acceptable, however, in this case the GMMG study office has to be consulted prior to study inclusion
* Patients with acute diffuse infiltrative pulmonary and/or pericardial disease
* Autoimmune haemolytic anaemia with positive indirect Coombs test or immune thrombocytopenia
* Platelet count < 75 x 109/l
* Haemoglobin ≤ 8.0 g/dl, unless related to MM
* Absolute neutrophil count (ANC) < 1.0 x 109/l (the use of colony stimulating factors within 14 days before the test is not allowed)
* Corrected serum calcium > 14 mg/dl (> 3.5 mmol/l)
* Unable or unwilling to undergo thromboprophylaxis
* Pregnancy and lactation
* Participant has any concurrent severe and/or uncontrolled medical condition or psychiatric disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study or that confounds the ability to interpret data from the study
* Subjects, who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
* Participation in other interventional clinical trials. This does not include long-term follow-up periods without active drug treatment of previous studies during the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Demonstration of superiority of iberdomide plus isatuximab compared to iberdomide with respect to bone marrow minimal residual disease (MRD). | 24 months after start of maintenance therapy
  The primary objective of this trial is to compare the two-year MRD negativity rate (sensitivity 2x10^-6 via next-generation flow cytometry [NGF]; from bone marrow aspirate) when treated with iberdomide plus isatuximab, with the MRD negativity after treatment with iberdomide only.

SECONDARY OUTCOMES:
Progression-free survival (PFS) from date of randomization. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  PFS, defined as time from randomization to disease progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Goldschmidt, Prof., Principal Investigator — University Hospital Heidelberg
Locations (69):
- Austria (5):
  - Universitätsklinikum Krems an der Donau, Krems
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Universitätsklinik für Innere Medizin III, Salzburg
  - Klinik Ottakring Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Germany (64):
  - Uniklinik RWTH Aachen, Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzelltransplantation, Aachen
  - Universitätsklinikum, Augsburg
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Charité, III. Medizinische Abteilung, Berlin
  - Vivantes Klinikum Neukölln, Klinik für Hämatologie und Onkologie, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Evangelisches Klinikum Bethel, Bielefeld
  - Johanniter Krankenhaus, Bonn
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum, Braunschweig
  - Klinikum Chemnitz, Chemnitz
  - Carl-Thiem-Klinikum Cottbus gGmbH, 2. Medizinische Klinik, Cottbus
  - Klinikum Darmstadt GmbH, Medizinische Klinik V, Darmstadt
  - Städtisches Klinikum, Dessau
  - St. Johannes Hospital Dortmund, Dortmund
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Marien Hospital Düsseldorf GmbH, Klinik für Onkologie, Hämatalogie und Palliativmedizin, Düsseldorf
  - St. Antonius-Hospital, Eschweiler
  - KEM I Evang. Kliniken Essen-Mitte gGmbH, Evangelisches Krankenhaus Essen-Werden gGmbH, Klinik für Hämatologie, Onkologie und Stammzelltransplantation, Essen
  - Malteser Krankenhaus, Flensburg
  - Universitätsklinikum Frankfurt, Frankfurt
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Greifswald, Greifswald
  - Katholisches Krankenhaus Hagen, Hagen
  - Universitätsklinikum Hamburg-Eppendorf, Zentrum für Onkologie, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Onkologische Schwerpunktpraxis, Heidelberg
  - Universitätsklinikum Heidelberg, Medizinische Klinik V, Heidelberg
  - SLK Kliniken Heilbronn, Medizinische Klinik III, Heilbronn
  - Universitätsklinikum des Saarlandes, Klinik für Innere Medizin 1, Homburg
  - Klinikum der Friedrich-Schiller-Universität Jena, Klinik für Innere Medizin II, Abteilung Hämatologie und internistische Onkologie, Jena
  - Westpfalz-Klinikum, Kaiserslautern
  - Klinikverbund Allgäu, Klinikum Kempten, Hämatologie / Onkologie, Kempten
  - Gemeinschaftsklinikum Mittelrhein Koblenz, Koblenz
  - Oncocare, Gemeinschaftspraxis für Hämatologie und Onkologie, Lebach
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität, Mainz
  - Universitätsklinikum Mannheim, III. Medizinische Klinik, Mannheim
  - Onkologie Praxis, Mannheim
  - Philipps-Universität Marburg Hämatologie/Onkologie, Marburg
  - Klinikum Hochsauerland, Meschede
  - Kliniken Maria Hilf, Mönchengladbach
  - Kliniken Ostalb, Mutlangen
  - Rotkreuzklinikum, München
  - Klinikum rechts der Isar der TU München, München
  - Klinikum Oldenburg, Oldenburg
  - Klinikum Osnabrück GmbH, Osnabrück
  - Brüderkrankenhaus St. Josef, Paderborn
  - Krankenhaus Barmherzige Brüder Regensburg, Klinik für Onkologie und Hämatologie, Regensburg
  - Universitätsklinikum Regensburg, Regensburg
  - Diakoneo Diak Klinikum, Schwäbisch Hall
  - ZAHO - Zentrum für ambulante Hämatologie und Onkologie, Siegburg
  - Onkologische Schwerpunktpraxis Speyer, Speyer
  - Klinikum der Landeshauptstadt Stuttgart - Katharinenhospital, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum, Ulm
  - Schwarzwald Baar Klinikum, Villingen-Schwenningen
  - University of Würzburg, Med. Klinik und Poliklinik II, Würzburg

IPD SHARING:
Plan to Share IPD: No